CLINICAL TRIAL: NCT03054883
Title: Observational Study for Patients With Newly Diagnosed Mantle Cell Lymphoma (MCL) Not Eligible for High-dose Therapy According to the Protocol Alternating R-CHOP and R-cytarabine Chemotherapy Regimen (3+3 Cycles)
Brief Title: Observational Study for Patients With Newly Diagnosed (MCL) Not Eligible for High-dose Therapy
Status: Completed | Type: Observational
Sponsor: Czech Lymphoma Study Group (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: Sponsor
Other Study IDs: CLSG-MCL-01
Record Dates: First submitted 2017-02-09; First posted 2017-02-16 (Actual); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle Cell Lymphoma; minimal residual disease; cytosine arabinoside
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Isolation of DNA from leukemized peripheral blood or infiltrated bone marrow will be used for set up of patient-specific primers for detection of minimal residual disease after induction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study aimed to analyze the effectiveness of treatment of patients with newly dg. mantle cell lymphoma not eligible for high-dose therapy and autologous stem cell transplantation. Scheme of treatment: alternating cycles of R-CHOP (rituximab, cyclophosphamide, hydroxydaunomycin, oncovin, prednison) and R-AraC (rituximab, cytarabin): R-CHOP / R-AraC / R-CHOP / R-AraC / R-CHOP / R-AraC. The study was proposed based on the previously published data in the younger patients, which demonstrated improved outcome after implementation of Ara-C into induction.

DETAILED DESCRIPTION:
This is an observational study considered for patients with mantle cell lymphoma meeting the basic inclusion criteria. The study will enrol patients who will be treated according to standard protocol used in the hematologic department. Scheme of treatment: alternating cycles of R-CHOP and R-AraC: R-CHOP / R-AraC / R-CHOP / R-AraC / R-CHOP / R-AraC.

Baseline procedures:

* CT or PET-CT (positron emission tomography with computed tomography)before starting treatment, after 3 cycles and at the end of treatment (after 6 cycles)
* bone marrow examination before therapy, after 3 cycles and after completion of induction
* maintenance rituximab based of standards of each centre

The study was proposed based on the previously published data in the younger patients, which demonstrated improved outcome after implementation of Ara-C into induction.

Primary objectives include response after induction by PET-CT and PFS (progression-free survival).

Secondary objectives include OS (overall survival), and prognostic significance of minimal residual disease detection after completion of induction

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of MCL (hematopathologic examination in the reference centre, with evidence of cyclin D1 or translocation t(11;14) )
* not eligible for high-dose therapy with autologous stem cell transplantation
* eligible for R-CHOP or R-COEP-based therapy
* signed informed consent form with the study and data processing

Exclusion Criteria:

* non compliance of a patient
* CNS (central nervous system) involvement with lymphoma
* ECOG (Eastern Cooperative Oncology Group) >3 or active uncontrolled comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly and/or comorbid patients with newly dg. mantle cell lymphoma not eligible for high-dose therapy and autologous stem cell transplantation, eligible for R-CHOP or R-COEP (rituximab, cyclophosphamide, oncovin, etoposide, prednison) based therapy.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Overall response | After induction for all patients, who can be evaluated; through study completion, an average of 1 year.
  PET-CT after induction, and bone marrow examination after induction

SECONDARY OUTCOMES:
Progression-free survival and overall survival | max. 4 years
  PFS will be calculated from initiation of therapy until lymphoma relapse / progression or death from any cause; OS will be calculated from initiation of therapy until death from any cause
Minimal residual disease (MRD) by PCR (polymerase chain reaction) after induction | After induction for all patients, who can be evaluated; through study completion, an average of 1 year.
  After completion of induction MRD will be evaluated by PCR in the peripheral blood and bone marrow in those patients with available disease markers, i.e. primers detecting the translocation t(11;14) or unique IgVH rearrangement.

CONTACTS AND LOCATIONS:
Overall Officials: Marek Trneny, prof.,PhD., Principal Investigator — Charles University General Hospital in Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klener P, Fronkova E, Belada D, Forsterova K, Pytlik R, Kalinova M, Simkovic M, Salek D, Mocikova H, Prochazka V, Blahovcova P, Janikova A, Markova J, Obr A, Berkova A, Kubinyi J, Vaskova M, Mejstrikova E, Campr V, Jaksa R, Kodet R, Michalova K, Trka J, Trneny M. Alternating R-CHOP and R-cytarabine is a safe and effective regimen for transplant-ineligible patients with a newly diagnosed mantle cell lymphoma. Hematol Oncol. 2018 Feb;36(1):110-115. doi: 10.1002/hon.2483. Epub 2017 Oct 30. PMID 29083050
- See also: Official Site of the Czech Lymphoma Study Group — http://www.lymphoma.cz